CLINICAL TRIAL: NCT00242944
Title: Japan Assessment of Pitavastatin and Atorvastatin in Acute Coronary Syndrome
Brief Title: Japan Assessment of Pitavastatin and Atorvastatin in Acute Coronary Syndrome (JAPAN-ACS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University (Other)
Collaborators: Yamaguchi University Hospital (Other); Juntendo University (Other)
Responsible Party: Principal Investigator, Takeshi Morimoto, Investigator, Kyoto University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H17-49
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Coronary Disease; Hypercholesterolemia
Keywords: Acute coronary syndrome; Hypercholesterolemia; Primary coronary intervention; Hydroxymethylglutaryl-CoA reductase inhibitors; coronary plaque; Angioplasty, Transluminal, Percutaneous Coronary; Ultrasonography, Interventional
MeSH Terms: conditions — Coronary Disease; Hypercholesterolemia; Acute Coronary Syndrome | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pitavastatin
  Interventions: Drug: Pitavastatin
- 2 (Active Comparator): Atorvastatin
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 4mg per day
  Arms: 1
Drug: Atorvastatin — Atorvastatin 20mg per day
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effects of pitavastatin and atorvastatin on coronary plaque volume in patients with acute coronary syndrome and to clarify the relationship between coronary plaque volume, serum lipids, and inflammation markers in order to determine the significance of intensive lipid lowering therapy in patients with acute coronary syndrome in Japan.

DETAILED DESCRIPTION:
Previous mega trials have demonstrated that lipid lowering therapy with HMG-CoA reductase inhibitors (statins) reduces the incidence of major cardiovascular events by one-third, thus, the benefit of lipid lowering therapy has been substantiated. Such a benefit is significant especially for patients with coronary heart disease (CHD). The third report of the National Cholesterol Education Program Adult Treatment Panel (NCEP ATP-III) has suggested the advantage of more intensive lipid lowering therapy with a goal of reducing LDL-C below 70 mg/dL for such patients categorized as very high risk. In Japan, Japan Atherosclerosis Society (JAS) Guidelines for Diagnosis and Treatment of Atherosclerotic Cardiovascular Diseases 2002 have recommended that an LDL-C goal for patients with coronary heart disease should be below 100 mg/dL. However, there is no satisfactory evidence yet for the need to lower LDL-C level less than the goal prescribed in Japan.

Recently, research on diagnosis of coronary plaque has shown significant advances. The REVERSAL study in patients with a history of CHD, by diagnosis with intravascular ultrasound, suggested that intensive lipid lowering therapy with atorvastatin (80 mg/day) was associated with no growth of plaque (-0.4% compared to baseline), versus therapy with pravastatin (40 mg/day) which showed a slight increase (2.7%) in plaque volume over 18 months. In Japan, the ESTABLISH study, a single center study, indicated that early intensive lipid lowering therapy with atorvastatin (20 mg/day) could induce a significant reduction in plaque volume in patients with acute coronary syndrome. However, this benefit has not been verified in multicenter trials in Japan. Further, no comparative investigation into the effect of various concomitant drugs on coronary plaque has been done.

Pitavastatin is a chemically synthesized statin in Japan which has been marketed since late 2003. Pitavastatin has an LDL-C lowering effect as strong as atorvastatin and also has a superior HDL-C elevating effect; meanwhile, the effect of pitavastatin on coronary plaque has not been reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients with written consent by their own volition after being provided sufficient explanation for their participation in this clinical trial
* Patients 20 years or older at the time of their consent
* Patients with hypercholesterolemia as defined by any of the following criteria:

  * TC >= 220 mg/dL;
  * LDL-C >= 140 mg/dL;
  * Cholesterol-lowering treatment is necessary in accordance with the investigator's judgement when LDL-C >= 100 mg/dL or TC >= 180 mg/dL.
* Patients who have been diagnosed with acute coronary syndrome
* Patients with successful percutaneous coronary intervention (PCI) by intravascular ultrasound (IVUS) guidance
* Patients having coronary plaques (>= 500 µm in thickness or 20% or more in % plaque) at >= 5 mm from the previously treated area in the same branch of coronary artery

Exclusion Criteria:

* Patients with bypass graft or in-stent restenosis at the site of PCI
* Patients who had received PCI on the lesion in the past where the evaluation of coronary plaque volume is planned
* Patients who had plaques in a non-culprit site and might receive PCI during the treatment period
* Patients receiving lipid-lowering drugs (statins, fibrates, probucol, nicotinic acid or cholesterol absorption inhibitors)
* Patients with familial hypercholesterolemia
* Patients with cardiogenic shock
* Patients receiving cyclosporine
* Patients with any allergy to pitavastatin or atorvastatin
* Patients with hepatobiliary disorders
* Pregnant women, women suspected of being pregnant, or lactating women
* Patients with renal disorders or undergoing dialysis
* Patients who are ineligible in the opinion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
plaque volume | one year

SECONDARY OUTCOMES:
total cholesterol (TC) | one year
low-density lipoprotein (LDL)-cholesterol (LDL-C) | one year
high-density lipoprotein (HDL)-cholesterol (HDL-C) | one year
HDL2-C | one year
HDL3-C | one year
remnant like particles-cholesterol (RLP-C) | one year
small dense LDL-C | one year
non-HDL-C | one year
LDL-C/HDL-C | one year
apolipoprotein AI (apoA-I) | one year
apoB | one year
apoE | one year
apoB/apoA-I | one year
malondialdehyde-modified LDL (MDA-LDL) | one year
phospholipids | one year
lipoprotein(a) [Lp(a)] | one year
high-sensitivity C-reactive protein (hs-CRP) | one year
pentraxin 3 | one year
leukocytes | one year
coronary plaque area at culprit region | one year
minimal lumen diameter (MLD) and percent (%) stenosis | one year
major adverse cardiac events (cardiac death, Q or non-Q myocardial infarction and target vessel revascularization) | one year
number of deaths from any cause | one year
frequency of adverse drug reactions | one year

CONTACTS AND LOCATIONS:
Overall Officials: Masunori Matsuzaki, MD, PhD, Study Chair — Professor of Medicine, Department of Cardiovascular Medicine, Yamaguchi University Graduate School of Medicine; Hiroyuki Daida, MD, Principal Investigator — Professor of Medicine, Department of Cardiovascular Medicine, Juntendo University School of Medicine; Takeshi Kimura, MD, Principal Investigator — Associate Professor of Medicine, Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (3):
- Japan (3):
  - Juntendo University School of Medicine, Bunkyo-ku, Tokyo
  - Yamaguchi University Graduate School of Medicine, Ube, Yamaguchi
  - Kyoto University Graduate School of Medicine, Kyoto

REFERENCES:
- [Background] Miyauchi K, Kimura T, Morimoto T, Nakagawa Y, Yamagishi M, Ozaki Y, Hiro T, Daida H, Matsuzaki M. Japan assessment of pitavastatin and atorvastatin in acute coronary syndrome (JAPAN-ACS): rationale and design. Circ J. 2006 Dec;70(12):1624-8. doi: 10.1253/circj.70.1624. PMID 17127811
- [Result] Hiro T, Kimura T, Morimoto T, Miyauchi K, Nakagawa Y, Yamagishi M, Ozaki Y, Kimura K, Saito S, Yamaguchi T, Daida H, Matsuzaki M; JAPAN-ACS Investigators. Effect of intensive statin therapy on regression of coronary atherosclerosis in patients with acute coronary syndrome: a multicenter randomized trial evaluated by volumetric intravascular ultrasound using pitavastatin versus atorvastatin (JAPAN-ACS [Japan assessment of pitavastatin and atorvastatin in acute coronary syndrome] study). J Am Coll Cardiol. 2009 Jul 21;54(4):293-302. doi: 10.1016/j.jacc.2009.04.033. PMID 19608026
- [Derived] Fukushima Y, Daida H, Morimoto T, Kasai T, Miyauchi K, Yamagishi S, Takeuchi M, Hiro T, Kimura T, Nakagawa Y, Yamagishi M, Ozaki Y, Matsuzaki M; JAPAN-ACS Investigators. Relationship between advanced glycation end products and plaque progression in patients with acute coronary syndrome: the JAPAN-ACS sub-study. Cardiovasc Diabetol. 2013 Jan 7;12:5. doi: 10.1186/1475-2840-12-5. PMID 23289728
- [Derived] Takashima H, Ozaki Y, Morimoto T, Kimura T, Hiro T, Miyauchi K, Nakagawa Y, Yamagishi M, Daida H, Mizuno T, Asai K, Kuroda Y, Kosaka T, Kuhara Y, Kurita A, Maeda K, Amano T, Matsuzaki M; JAPAN-ACS Investigators. Clustering of metabolic syndrome components attenuates coronary plaque regression during intensive statin therapy in patients with acute coronary syndrome: the JAPAN-ACS subanalysis study. Circ J. 2012;76(12):2840-7. doi: 10.1253/circj.cj-11-1495. Epub 2012 Sep 7. PMID 22972364
- [Derived] Ohashi T, Shibata R, Morimoto T, Kanashiro M, Ishii H, Ichimiya S, Hiro T, Miyauchi K, Nakagawa Y, Yamagishi M, Ozaki Y, Kimura T, Daida H, Murohara T, Matsuzaki M. Correlation between circulating adiponectin levels and coronary plaque regression during aggressive lipid-lowering therapy in patients with acute coronary syndrome: subgroup analysis of JAPAN-ACS study. Atherosclerosis. 2010 Sep;212(1):237-42. doi: 10.1016/j.atherosclerosis.2010.05.005. Epub 2010 May 11. PMID 20684825
- [Derived] Hiro T, Kimura T, Morimoto T, Miyauchi K, Nakagawa Y, Yamagishi M, Ozaki Y, Kimura K, Saito S, Yamaguchi T, Daida H, Matsuzaki M; JAPAN-ACS Investigators. Diabetes mellitus is a major negative determinant of coronary plaque regression during statin therapy in patients with acute coronary syndrome--serial intravascular ultrasound observations from the Japan Assessment of Pitavastatin and Atorvastatin in Acute Coronary Syndrome Trial (the JAPAN-ACS Trial). Circ J. 2010 Jun;74(6):1165-74. doi: 10.1253/circj.cj-09-0766. Epub 2010 May 12. PMID 20467151